CLINICAL TRIAL: NCT07271589
Title: Biological and Clinical Underpinnings of Postoperative Pain - Mastectomy (BAC-UPP 1 Study)
Brief Title: Biological and Clinical Underpinnings of Postoperative Pain - Mastectomy
Acronym: BAC-UPP 1
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Demario Overstreet, Assistant Professor of Surgery, University of Alabama at Birmingham
Other Study IDs: IBR-300015322; 1R35GM159908-01 (NIH)
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Mastectomy
Keywords: Mastectomy; breast surgery; nociception; acute pain; chronic pain
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Specimen Collection: The following biomarkers: (proinflammatory) Fibrinogen, Serum Amyloid A, interleukin-1 alpha (IL-1α), 1IL-1β, IL-6, Tumor necrosis factor-alpha (TNF-α), and (Anti-inflammatory) Vitamin D, IL4, IL10, IFN-a will be determined by implementing the Meso Scale Discovery, which is an enzyme-linked immunosorbent assay (ELISA) that employs electrochemiluminescence to identify specific binding events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Surgery/Mastectomy Patients

SUMMARY:
Persistent pain after mastectomy remains a significant clinical challenge that can delay recovery, reduce quality of life, and increase long-term healthcare burden. The goal of this study is to gain a deeper understanding of the biological and clinical factors that influence pain severity after mastectomy and contribute to the transition from acute to chronic postoperative pain. Guided by a biopsychosocial framework, this research will address the following aims:

1. We will use standardized experimental pain testing before surgery to evaluate how patients respond to different types of controlled sensory stimuli. These responses may help predict who is more likely to experience severe or prolonged pain after surgery.
2. We will analyze blood samples collected before and after surgery to measure markers of inflammation and other biological responses. These data will help us explore how the body's immune and hormonal systems relate to pain severity in both the short- and longer-term recovery phases.
3. We will assess psychological and clinical factors, such as emotional health, coping style, household income, and life stressors, to understand how they contribute to patients' pain experiences throughout recovery.
4. We will examine whether routinely collected demographic and clinical characteristics can help identify patients at greater risk of experiencing higher levels of pain after surgery. This approach will allow us to better understand which patients may benefit from more tailored perioperative pain management strategies.

DETAILED DESCRIPTION:
The overarching goal of this study is to elucidate the biological, psychological, and clinical factors that are responsible for pain trajectories following mastectomy. Using a biopsychosocial framework, we aim to identify modifiable risk and protective mechanisms that could inform the development of targeted interventions to prevent chronic postsurgical pain.

Aim 1: Characterize individual differences in pain processing using standardized experimental pain testing.

Participants will complete a battery of quantitative sensory testing (QST) measures preoperatively to assess their sensitivity to mechanical, thermal, and pressure-based stimuli. These standardized tests capture individual differences in nociceptive and central pain modulation. By linking preoperative pain sensitivity profiles to postoperative pain intensity and duration, we will determine whether QST-derived measures can serve as early predictors of maladaptive pain trajectories.

Aim 2: Examine biological and inflammatory mechanisms underlying postoperative pain persistence.

Peripheral blood samples will be collected at multiple time points before and after surgery to quantify circulating markers of inflammation (e.g., IL-6, CRP), neuroendocrine function (e.g., oxytocin, vasopressin), and immune regulation. These biomarkers will be analyzed in relation to clinical pain outcomes to identify biological signatures associated with resilience versus vulnerability to chronic pain. This aim will provide mechanistic insight into how systemic physiological responses to surgery contribute to prolonged nociceptive signaling.

Aim 3: Assess psychosocial determinants of pain and recovery.

We will evaluate key psychological and social-contextual variables, including emotional health, coping style, catastrophizing, optimism, perceived stress, and socioeconomic indicators-to determine how these factors influence postoperative pain experiences and recovery. This comprehensive assessment will clarify how psychological resilience and environmental stressors interact with biological processes to shape individual pain outcomes.

Aim 4: Develop a multidimensional risk model integrating demographic, clinical, and mechanistic predictors.

Using routinely collected demographic and perioperative data (e.g., age, sex, race, comorbidities, analgesic use, surgical approach), combined with the experimental, biological, and psychosocial measures from Aims 1-3, we will construct an integrative predictive model of postoperative pain outcomes. This approach will allow us to identify distinct risk phenotypes and generate clinically actionable profiles for early identification of patients most likely to benefit from personalized perioperative pain management strategies.

Together, these efforts will advance our understanding of how biological, psychological, and contextual factors jointly influence pain recovery after surgery, with the long-term goal of informing precision pain medicine and improving postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Participants scheduled for breast surgery/mastectomy ; 2) age between 18-65; 3) understanding of verbal and written English.

Exclusion Criteria:

* 1) concurrent medical conditions that could confound the interpretation of the data; 2) HIV positive diagnosis; 3) cardiovascular or pulmonary disease; 4) systemic rheumatoid disease; 5) uncontrolled hypertension (i.e. SBP/DBP of > 150/95); 6) current illness accompanied by fever (body temperature >38 °C); 7) any other chronic pain condition; 8) conditions resulting in altered nerve sensation; 9) hospitalization due to psychiatric illness within the last 6 months; 10) poorly controlled diabetes; 11) history of stroke; 12) history of seizures; 13) circulatory disorders such AS Raynauds' disease 14) history of drug or alcohol abuse.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Pain after Mastectomy (Using Brief Pain Inventory - Short Form) | 12 weeks after surgery
  Pain measured 3 months following mastectomy
  The BPI-SF is a multidimensional pain scale used to assess self-reported pain severity and its interference with daily functioning. The questionnaire is composed of four items asking about pain severity (worst pain, least pain, average pain, and pain right now) over the past 24 h. Additionally, seven items assess the degree to which pain interferes with functioning in the following domains: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Each item is scored from 0 (no pain or does not interfere) to 10 (worst imaginable pain or completely interferes). Higher scores suggest greater pain severity and pain interference. The BPI-SF is a well validated chronic pain questionnaire that has previously been used in samples with cLBP.
Acute Pain after Surgery (using Brief Pain Inventory- Short Form) | 48 hours after surgery
  Pain rating 48 hours after surgery using Brief Pain Questionnaire
  The BPI-SF is a multidimensional pain scale used to assess self-reported pain severity and its interference with daily functioning. The questionnaire is composed of four items asking about pain severity (worst pain, least pain, average pain, and pain right now) over the past 24 h. Additionally, seven items assess the degree to which pain interferes with functioning in the following domains: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Each item is scored from 0 (no pain or does not interfere) to 10 (worst imaginable pain or completely interferes). Higher scores suggest greater pain severity and pain interference. The BPI-SF is a well validated chronic pain questionnaire that has previously been used in samples with cLBP.

IPD SHARING:
Plan to Share IPD: Yes
de-identified QST data, biomarkers, survey responses, demographics
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available 6 months after publication of primary results
Access Criteria: This data/information will be made available via email request

REFERENCES:
- [Background] Overstreet DS, Strath LJ, Sorge RE, Thomas PA, He J, Wiggins AM, Hobson J, Long DL, Meints SM, Aroke EN, Goodin BR. Race-specific associations: inflammatory mediators and chronic low back pain. Pain. 2024 Jul 1;165(7):1513-1522. doi: 10.1097/j.pain.0000000000003154. Epub 2024 Feb 6. PMID 38323608
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Horn R, Hendrix JM, Kramer J. Postoperative Pain Control. 2024 Jan 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK544298/ PMID 31335018
- [Background] Dobson GP. Trauma of major surgery: A global problem that is not going away. Int J Surg. 2020 Sep;81:47-54. doi: 10.1016/j.ijsu.2020.07.017. Epub 2020 Jul 29. PMID 32738546
- [Background] Small C, Laycock H. Acute postoperative pain management. Br J Surg. 2020 Jan;107(2):e70-e80. doi: 10.1002/bjs.11477. PMID 31903595
- [Background] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Background] Bruce J, Quinlan J. Chronic Post Surgical Pain. Rev Pain. 2011 Sep;5(3):23-9. doi: 10.1177/204946371100500306. PMID 26526062